CLINICAL TRIAL: NCT01135199
Title: Safety and Efficacy of Pomalidomide in the Treatment of Refractory Cough in Patients With Idiopathic Pulmonary Fibrosis (IPF): A Pilot Study
Brief Title: Pomalidomide for Cough in Patients With Idiopathic Pulmonary Fibrosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA did not accept sponsor's animal toxicology data to support proposed dosing.
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Paul Mohabir, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-05302008-1189
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): Open label
  Interventions: Drug: pomalidomide (CC-4047

INTERVENTIONS:
Drug: pomalidomide (CC-4047

SUMMARY:
The purpose of this study is to determine the safety and efficacy of pomalidomide over a 12 week duration in the treatment of chronic cough in patients with IPF as measured by a Cough Symptom Diary, Visual Analogue Scale for Cough Severity, Leicester Cough Questionnaire, St. George Respiratory Questionnaire, Cough-Specific Quality-of-Life Questionnaire, and adverse event reporting. There will be an option open to participants, who respond to treatment by meeting pre-determined criteria, to remain in the study for an additional 9 months or for a total of 54 weeks.

DETAILED DESCRIPTION:
Chronic cough is one of the most debilitating symptoms in patients with IPF. It is estimated that over 80% of patients with IPF experience clinically significant cough. The impact of chronic cough on QOL includes fatigue, embarrassment, anxiety, sleep disturbance, hoarseness, incontinence, dizziness, vomiting, rib fractures, and severe dyspnea. There is also some evidence that chronic cough may contribute to increased airway inflammation. In IPF patients, significant oxygen desaturation often accompanies coughing episodes leading to increased dyspnea, anxiety, and panic. Studies examining alternative therapeutic agents for cough in IPF patients are scarce. Cough in patients with IPF is typically refractory to traditional antitussive agents or corticosteroids.

Unfortunately, the side effects of corticosteroids combined with their lack of efficacy in prevention of disease progression in IPF makes this a less desired treatment option.

Although opiates can be effective in controlling cough, issues of sedation, respiratory depression and narcotic dependence are significant.

This is an open label, safety and efficacy pilot study of pomalidomide in 20 patients with IPF. This study will determine both the tolerability and feasibility of pomalidomide for the treatment of cough in this patient population.

Eligible patients will be selected from our Interstitial Lung Disease Clinic database which consists of patients with ILD seen in our clinic since about 2004 who have signed informed consent (previously approved by our Administrative Panel on Human Subjects in Medical Research, protocol 14054). Those patients with IPF who describe the severity of their cough as decreasing, or adversely affecting, their quality of life will be invited to participate in the study.

SCREENING VISIT During this visit, the study will be fully reviewed with the patient, who will already have received the consent form and discussed it by phone, or at a previous clinic visit with the study coordinator and possibly the PI or Sub PI. At this visit the pt. will undergo Informed Consent, bloodwork including Chem Panel with LFTs, CBC, History and Physical Exam - MD, Vital Signs, Spirometry without Bronchodilator, Diffusion Capacity, 6 Minute Walk, EKG, Adverse Events, Cough Visual Analog Scale (VAS), Leicester Cough Questionaire (LCQ), Cough-Specific Quality-of-Life Questionnaire (CQLQ),St. George Respiratory Questionnaire (SGRQ), and dispensation of the Cough Symptom Diary (CSD).

If the patient continues to meet eligibility criteria, current cough suppressive agents will be discontinued from days 1-14.

STUDY DAY 1, VISIT 1 History and Physical Exam - MD, Vital Signs, Adverse Events, Cough Visual Analog Scale, LCQ, CQLQ and the SGRQ. The patient will then be given a 30 day supply of 2mg capsules of pomalidomide with written instructions on dosing and instructions to call the study center with any adverse reactions.

WEEK 1, Visit 2 Pt. will come to study site for safety labs, and assessment of adverse events and any changes in medications.

WEEK 2, VISIT 3 The patient will return to the clinic to be assessed for potential adverse reactions and to have safety laboratory work done.

WEEKS 4, 8, and 12 (Visits 4, 6, and 8) The participant will return to the study center and undergo physical exam, vital signs, assessment of adverse events, and self-completion of the VAS, LCQ, and the CQLQ. Every two weeks (Visits 2, 4, and 6) the patient will also undergo safety laboratory testing which can either be done at Stanford or at a local lab. As part of routine care, we will obtain spirometry and 6MWT at the start and end of study. If there are abnormalities in the patient's labs at week 2 we will either withdraw the patient from the study or down-titrate their dose depending on the severity of lab abnormality.

A 30 day supply of 2mg capsules of pomalidomide will be dispensed at Week 4 and 8.

The patient will undergo a 2 week taper to 1 mg/day of study drug at week 12 to off drug by wk. 14, and will have a return follow up visit at week 18 for assessment of adverse events, history and physical exam, lab work including pregnancy test, and completion of all four questionnaires.

Patients responding by meeting the established minimally clinically important difference for the CQLQ as well as having demonstrated safety tolerance by laboratory tests and physician exam and who wish to remain in the study may do so for an additional 9 months at the discretion of the Protocol Director. These participants will not undergo taper at week 12 and will be re-supplied on a monthly basis until week 48 at which time they will taper to off drug over 2 weeks.

The Visit Schedule for the extension study is the same as the initial 3 months with the exception that safety laboratory blood work is done monthly instead of every two weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. >18 and < 75 years old at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Have a diagnosis of Idiopathic Pulmonary Fibrosis in accordance to American Thoracic Society guidelines.
5. Persistent cough:

   • as defined by a cough that adversely affects the patient's quality of life and has been present for at least 3 months.
6. Laboratory test results within these ranges:

   * Absolute neutrophil count >2 x 103/ul
   * Platelet count >100,000 /mm³
   * Serum creatinine < 2.0 mg/dL
   * Total bilirubin < 1.5 mg/dL
7. Diffusion capacity > 25%predicted
8. Forced vital capacity <80% predicted • AST (SGOT) and ALT (SGPT) < 2 x ULN

8. Able to take aspirin (81 or 325 mg) daily as prophylactic anti-coagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Females of child-bearing potential defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental drug or therapy within 28 days of baseline.
5. Known hypersensitivity to thalidomide or lenalidomide.
6. Any prior use of thalidomide, lenalidomide or pomalidomide (CC-4047).
7. Known positive for HIV or infectious hepatitis, type A, B or C.
8. History of deep venous thrombosis
9. History of pulmonary embolism
10. Use of the following anti-tussive agents must be discontinued 14 days prior to their baseline visit. -

1. prednisone 2. narcotic anti-tussives 3. baclofen 4. neurontin 11. Treatment for infection or acute exacerbation within past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: Cough related QOL as measured by Cough-Specific Quality of LIfe instrument (CQLQ) | 12 weeks

SECONDARY OUTCOMES:
Outcome Measure: Cough severity as measured by Leicester Cough Questionnaire (LCQ), Visual Analog Scale (VAS), St. George Respiratory Questionnaire (SGRQ) | 12 wks

CONTACTS AND LOCATIONS:
Overall Officials: Glenn D. Rosen, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Horton MR, Danoff SK, Lechtzin N. Thalidomide inhibits the intractable cough of idiopathic pulmonary fibrosis. Thorax. 2008 Aug;63(8):749. doi: 10.1136/thx.2008.098699. No abstract available. PMID 18663075